CLINICAL TRIAL: NCT06244355
Title: Studies of Phenotypic and Functional Characteristics of Circulating Neutrophil Subpopulations in Patients With Lung Cancer Undergoing Treatment
Brief Title: Studies of Phenotypic and Functional Characteristics of Circulating Neutrophil Subpopulations in Patients With Lung Cancer
Acronym: PNN-CP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220335; 2021-A01939-32 (Other: France : ANSM)
Record Dates: First submitted 2023-10-27; First posted 2024-02-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Neutrophils; neutrophil subsets; Advanced lung cancer; biomarkers; PD-1 immunotherapy; Chronic inflammation; Phenotypic modulation; Spectral cytometry
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Lung cancer: Metastatic, with complete mutational status, without anterior treatment
  Interventions: Other: Extra blood tubes
- Chronic obstructive pulmonary disease (COPD): Diagnosis of post-smoking COPD (without diagnosis of CP)
  Interventions: Other: Extra blood tubes
- Healthy volunteers: Healthy volunteers (based on biological and clinical data already available from the partner)
  Interventions: Other: Extra blood tubes

INTERVENTIONS:
Other: Extra blood tubes — Extra blood tubes

SUMMARY:
The objective is to study the phenotypic, functional and metabolomic characteristics of neutrophils circulating subpopulations in lung cancer patients, and to compare them to a control group of healthy volunteers. A blood sample will be taken before the first treatment session for the lung cancer patient and a second blood sample will be taken during the first evaluation visit.

The investigators hypothesize that there may be different circulating neutrophil subpopulations in patients with metastatic non-small cell lung cancer (NSCLC) involved in tumor progression and resistance to immunotherapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) have been shown to be effective in metastatic lung cancer. Unfortunately, 80% of patients do not respond and show rapid disease progression. Identifying predictive biomarkers of response is essential for early adaptation of management. Circulating lymphocytes and neutrophils represent a biomarker (NLR), predictive of immunotherapy response, in particular via the measurement of the neutrophils /lymphocyte ratio. Some preclinical work suggests a role for circulating neutrophil subpopulations like MDSC (myeloid derived suppressor cells) in ICI resistance. Certain circulating neutrophil subpopulations are thought to promote tumor progression, angiogenesis and metastasis with immunosuppressive activity. Identifying these pro-tumor subpopulations could predict the response to ICI and could be a potential therapeutic target. Our goal is to characterize the circulating neutrophil subpopulations of lung cancer patients and correlate these characteristics with response and survival phenotypically and functionally.

ELIGIBILITY:
Inclusion Criteria common to lung cancer and COPD patients :

* Age ≥ 18 years,
* male or female,
* affiliated with a Health Insurance,

Inclusion Criteria for lung cancer patients :

- Diagnosis of metastatic stage lung cancer with mutation status, naïve treatment

Inclusion Criteria for COPD patients :

- Diagnosis of COPD post-smoking

Exclusion Criteria:

* Tuberculosis or other acute or chronic bacterial infections
* Chronic progressive viral infections (Hepatitis B and C, HIV)
* Previous or ongoing chemotherapy
* Impossibility of giving the subject informed information.
* Opposition to the research.
* Participation in another research study with an exclusion period still in progress at pre-inclusion (possible inclusion in an observational study)
* Vulnerable individual (pregnant, parturient or breastfeeding woman), persons under guardianship or curatorship, or deprived of liberty by a judicial or administrative decision)
* Patients benefiting from the AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic lung cancer, without anterior treatment. Inclusion during a consultation or hospitalization by a pneumologist or oncologist in the thoracic oncology unit during care.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of a subpopulation of circulating neutrophils | Through study completion, an average of 3 years
  Presence of a subpopulation of circulating neutrophils in patients with lung cancer (absent in healthy volunteers and COPD patients) with phenotypic CD45+, CD15+, CD16+, CD62L-, LOX1+ and functional immunosuppressive characteristics.

SECONDARY OUTCOMES:
Demographic characteristics | Day 1
  Demographic characteristics : age, sex and smoking
Performans status | Day 1
  Somatic characteristics
Stage | Day 1
  Somatic characteristics
Histologic type | Day 1
  Histologic characteristics
Mutation status | Day 1
  Molecular characteristics
Clinical assessment | Up to the end of participation, between month 3 and month 4
  Progression free survival (defined as the time between the start of treatment and the date of first observation of clinical or CT progression (irRECIST1.1 criterion) or death)
irRECIST 1.1 response | Up to the end of participation, between month 3 and month 4
  CT scan to evaluate progression free survival (defined as the time between the start of treatment and the date of first observation of clinical or CT progression (irRECIST1.1 criterion) or death)
Death | Up to the end of participation, between month 3 and month 4
  Progression free survival (defined as the time between the start of treatment and the date of first observation of clinical or CT progression (irRECIST1.1 criterion) or death)
Mortality | Up to the end of participation, between month 3 and month 4
  Overall survival (defined as the time from treatment diagnosis to the date of death).

CONTACTS AND LOCATIONS:
Overall Officials: Marie WISLEZ, Pr, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP) - Cochin Hospital - Pneumology unit, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No